CLINICAL TRIAL: NCT07060196
Title: The Impact of Artificial Lighting on the Visual Capacity of Patients With Age-Related Macular Degeneration.
Acronym: ADLs AMD
Status: Not yet recruiting | Type: Observational
Sponsor: Democritus University of Thrace (Other)
Responsible Party: Principal Investigator, Georgios Labiris, Associate Professor of Ophthalmology, Democritus University of Thrace
Other Study IDs: ES20/Th62/23-11-2023
Record Dates: First submitted 2025-06-19; First posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: AMD - Age-Related Macular Degeneration
Keywords: AMD; artificial lighting; ADLs
MeSH Terms: conditions — Macular Degeneration | interventions — Tomography, Optical Coherence; Optical Imaging

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control Group: Healthy controls
  Interventions: Diagnostic Test: Distant Visual Acuity; Diagnostic Test: Optical Coherence Tomography; Diagnostic Test: Optical Coherence Tomography Angiography
- AMD Patients: Patients with AMD stage 9 in both eyes.
  Interventions: Diagnostic Test: Distant Visual Acuity; Diagnostic Test: Optical Coherence Tomography; Diagnostic Test: Optical Coherence Tomography Angiography; Diagnostic Test: Autofluorescence imaging

INTERVENTIONS:
Diagnostic Test: Distant Visual Acuity — Distant Visual acuity of all participants using DDART web-application monocularly in both eyes.
Diagnostic Test: Optical Coherence Tomography — Optical Coherence Tomography of the macula will be performed to all patients.
Diagnostic Test: Optical Coherence Tomography Angiography — Optical Coherence Tomography Angiography of the macula will be performed to all patients.
Diagnostic Test: Autofluorescence imaging — Autofluorescence imaging using fundus camera for AMD staging.
  Groups: AMD Patients

SUMMARY:
Age-related macular degeneration (AMD) is the leading cause of irreversible vision loss in the elderly worldwide. The dry, non-exudative form of the disease, although more common, is associated with gradual and significant decline in functional vision. Despite advancements in diagnostic and therapeutic approaches, a targeted intervention that improves the daily functionality of these patients is still lacking. One critical, yet often overlooked, factor that affects daily performance is lighting conditions.

This study aims to objectively assess the impact of different lighting intensity levels on patients with advanced dry AMD during the execution of everyday activities. A total of 60 individuals will be evaluated (30 healthy controls over 60 years of age and 30 patients with clinically diagnosed advanced AMD, according to NICE and AREDS criteria). Participants will undergo ophthalmological assessment (visual acuity, contrast sensitivity, OCT/OCTA, autofluorescence), and their performance on five functional tasks (mobility, object grasping, sit-to-stand transition, obstacle avoidance, and hanging clothes) will be evaluated under eight lighting levels (20-300 lux) at a constant color temperature (4000K), in a specially designed laboratory equipped with motion and eye-tracking systems.

The primary endpoint is overall performance, based on task completion time and errors, expressed on a custom performance scale (0-100). Secondary data include changes in pupil size as an indicator of visual adaptation. The study aims to determine the optimal lighting range that maximizes functional vision and improves the quality of life for patients with AMD.

DETAILED DESCRIPTION:
Introduction Aging is associated with an increased prevalence of neurodegenerative disorders and leads to irreversible changes in both humans and animal models. The retina, a layer of neural tissue that lines the interior of the eyeball, is exposed to various harmful and stressful environmental factors, including age-related changes, which affect its function. Age-related macular degeneration (AMD) is the leading cause of visual decline and blindness worldwide in individuals aged 65 years and older. The number of patients suffering from AMD is expected to increase significantly in the coming decades. AMD primarily affects the macular region of the retina, which is responsible for central vision. It has a significant impact on patients' lives due to the loss of sharp and color vision, interfering with daily activities such as recognizing faces and reading.

To date, there is no proven treatment that slows or prevents the progression of advanced AMD. Laser photocoagulation and photodynamic therapy reduce the risk of moderate or severe vision loss in some individuals with the neovascular form of the disease. Other medical and surgical interventions are under investigation, but none have been shown to be effective. Identifying the exact pathophysiological mechanisms of AMD remains challenging. However, clinico-pathological observations and epidemiological studies have provided valuable insights into potential pathways involved in AMD development. AMD is generally classified into two forms: non-exudative (dry or atrophic) and exudative (wet).

Exudative AMD is characterized by the development of choroidal neovascularization (CNV), i.e., fibrovascular tissue that grows from the choriocapillaris, penetrates through breaks in Bruch's membrane into the sub-retinal pigment epithelium (RPE) space, and then under the neurosensory retina. Dry AMD involves dysfunction in the RPE-Bruch's membrane-choriocapillaris complex, resulting in lesions such as drusen (small, yellow-white deposits located mainly in the macular area), focal pigment clumping, and RPE atrophy. The most severe atrophic lesion observed in AMD is geographic atrophy, characterized by a well-demarcated round or oval area of depigmentation or clear absence of RPE cells.

The wet form of AMD represents less than 10% of cases but can lead to severe complications if untreated. The latest approach in CNV treatment includes intravitreal injections of anti-angiogenic agents. Vascular Endothelial Growth Factor (VEGF) plays a key role in angiogenesis and in the development of all forms of wet AMD, regardless of angiographic appearance, and increases vascular permeability. Anti-VEGF drugs aim to inhibit VEGF activity, thereby suppressing neovascular growth and reducing vascular leakage. However, this therapy merely delays disease progression. Thus, there is a need for novel preventive and therapeutic strategies targeting AMD.

One factor influencing AMD patients' ability to perform daily activities is lighting conditions. According to current literature, the ideal lighting conditions for AMD patients have not yet been thoroughly studied. Recently, our research team published a pioneering mathematical model to determine optimal lighting intensity in phakic and pseudophakic patients. Identifying optimal lighting for AMD patients could greatly enhance their quality of life.

It is also known that some individuals overestimate or underestimate their functional daily abilities based on self-assessed visual performance using questionnaires. Moreover, visual acuity alone is insufficient to provide a comprehensive assessment of patients' visual capacity. Ideally, any functional impairment should be objectively and realistically evaluated for each patient, either at home or in their work environment, by carefully assessing their performance in specific daily tasks.

Various activities have been developed to assess distance, as well as near and intermediate visual abilities. Mobility has been assessed in individuals with glaucoma using a specific framework of daily activities, and near/intermediate vision tasks have been evaluated in AMD patients. In contrast, performance in individuals with presbyopia and in those who have undergone presbyopia-correcting surgery has been evaluated using a different activity framework under stable or variable lighting conditions to determine optimal illumination levels.

Purpose The aim of this study is to evaluate the performance of patients with advanced-stage dry AMD in daily activities under different lighting conditions.

Method

This is a prospective observational comparative study involving a total of 60 participants, divided into two groups:

Healthy controls over the age of 60

Patients with bilateral diagnosed advanced AMD (according to the UK's National Institute for Health and Care Excellence-NICE-or AREDS 9-step classification), fulfilling at least one of the following criteria:

i) Geographic atrophy of the macula ii) Best-corrected visual acuity in the affected eye <6/18 or logMAR >0.4 with dense/confluent drusen, advanced RPE changes, or vitelliform lesions iii) Fibrous scar iv) RPE tear v) Atrophy (absence/thinning of RPE and/or retina) vi) Cystoid degeneration (persistent intraretinal fluid or tubular structures unresponsive to therapy)

All participants will undergo a clinical evaluation at the Ophthalmology Outpatient Clinic and the Gait Analysis Laboratory of the University General Hospital of Evros. Initial assessments will include best-corrected monocular visual acuity using the validated DDiVAT chart and contrast sensitivity using the Pelli-Robson chart. Diagnostic evaluations will include macular optical coherence tomography (OCT), OCT angiography (OCT-A), and fundus autofluorescence imaging for AMD staging. All examinations will be conducted in accordance with standard clinical practice, without any interventional medical procedures.

Following clinical evaluation, participants will perform five daily activities under eight different lighting intensities (20, 50, 100, 125, 150, 200, 250, and 300 lux), with fixed light temperature (4000K). The performance will be assessed at the Gait Analysis Laboratory, which features a custom lighting setup of four adjustable light fixtures, installed based on a professional lighting design study.

The lab is equipped with an infrared motion-detection camera system, which, through special body-mounted reflectors, captures full-body movement, task duration, and motion fluidity in real time.

Additionally, the setup includes eye-tracking glasses, capable of measuring pupil size, blink rate, and saccadic eye movements. All devices are controlled by integrated software that extracts the data mentioned above. This system will be used to evaluate patients' performance in daily tasks under each lighting condition.

Daily Activities

Mobility: Patients walk a set distance along a corridor with grey obstacles at their self-selected pace.

Reach and grasp tasks: A white table is divided into 9 sections. Three small (24 mm), three medium (55 mm), and three large (73 mm) objects are randomly placed. Participants are asked to locate a specific object and place it on a marked black cross at a designated spot.

Sit-to-stand and stand-to-sit: Patients transition between two chairs placed opposite each other, repeating the sequence three times as fast as possible.

Overhead obstacle avoidance: Patients pass under a stretched rope placed at 1.5 m height.

Clothesline task: Patients pick up four differently colored garments from a basket and hang them on a fixed clothesline using clothespins.

Primary Outcome Activity Scores: Each participant's activity score will be calculated based on task completion time and errors. Errors will incur time penalties. A total completion time will be derived for each activity under each lighting condition. A custom scoring scale from 0 (lowest) to 100 (highest) will be developed. Each participant's performance score will be generated from this scale, determining the optimal lighting condition for AMD patients.

Secondary Outcome Pupil Size: The behavior of patients' pupil sizes under different lighting conditions will be assessed to correlate pupil response with light intensity.

Statistical Analysis An a priori power analysis was conducted. For an effect size of 0.17 of the activity score, 26 participants will be required in each study group to achieve a power of 0.8 at a significance level of 0.05. The normality of measurement data will be assessed using the Shapiro-Wilk test. Normally distributed data will be analyzed with the t-test. Non-normally distributed data will be analyzed with the Mann-Whitney U test. p-values < 0.05 will be considered statistically significant. All statistical analyses will be performed using the Medcalc statistical software (Medcalc Software, Mariakerke, Belgium).

ELIGIBILITY:
Inclusion Criteria:

* Healthy controls over the age of 60.
* Diagnosis of bilateral dry age-related macular degeneration (AMD).

Exclusion Criteria:

* Patients with other ocular conditions such as high myopia, glaucoma, clinically significant diabetic retinopathy, and other diseases that may confound the evaluation of ocular outcome measurements.
* Patients who have undergone intraocular surgeries, except for uncomplicated cataract extraction surgery performed at least 3 months prior to their inclusion in the study.
* Individuals with systemic diseases, including oxalate kidney stones, Wilson's disease, hemochromatosis, lung cancer, or other illnesses associated with poor five-year survival.
* Patients with binocular best-corrected distance visual acuity less than or equal to hand motion perception.
* Patients with neurological, orthopedic, or psychiatric disorders that prevent them from completing the activities or conditions that may affect their performance.

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * Healthy controls over the age of 60
  * Patients with bilateral diagnosed advanced AMD (according to the UK's National Institute for Health and Care Excellence-NICE-or AREDS 9-step classification [13]), fulfilling at least one of the following criteria:
    i) Geographic atrophy of the macula ii) Best-corrected visual acuity in the affected eye <6/18 or logMAR >0.4 with dense/confluent drusen, advanced RPE changes, or vitelliform lesions iii) Fibrous scar iv) RPE tear v) Atrophy (absence/thinning of RPE and/or retina) vi) Cystoid degeneration (persistent intraretinal fluid or tubular structures unresponsive to therapy)
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2025-06-30 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
ADL score | On the same day as clinical evaluation, approximately 2-4 hours following baseline assessments.
  Each participant's activity score will be calculated based on task completion time and errors. Errors will incur time penalties. A total completion time will be derived for each activity under each lighting condition. A custom scoring scale from 0 (lowest) to 100 (highest) will be developed. Each participant's performance score will be generated from this scale, determining the optimal lighting condition for AMD patients.

SECONDARY OUTCOMES:
Pupil Size | On the same day as clinical evaluation, approximately 2-4 hours following baseline assessments.
  The behavior of patients' pupil sizes under different lighting conditions will be assessed to correlate pupil response with light intensity.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Alexandroupolis, Alexandroupoli, Greece

IPD SHARING:
Plan to Share IPD: No